CLINICAL TRIAL: NCT00523055
Title: Ultrasound-guided Supraclavicular Brachial Plexus Blockade: A Pharmacokinetic Study of Lidocaine and Adrenaline
Brief Title: Ultrasound-guided Supraclavicular Brachial Plexus Blockade
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical volume of patients for recruitment stopped.
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2007:078
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2011-04

CONDITIONS: Pain
Keywords: Pain; Brachial Plexus Anesthesia; Plasma Lidocaine Levels; Ultrasound
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lidocaine — Lidocaine, 5 mg/kg, via needle placed adjacent to brachial plexus with ultrasound, dosing separated by 1 week, 2 doses in total, one block will contain 5 mcg/kg of adrenaline

SUMMARY:
Pain Clinic patients undergoing physiotherapy for rehabilitation often have arm freezing performed. The quality of physiotherapy is felt to be superior with good pain control. The quality of the freezing is felt to be better when it is done with ultrasound guidance. We are able to use less drug to achieve the same result. For this reason, we are doing a study to look at the level of freezing drug that accumulates in the body. We feel that the drug levels will be significantly different. We also feel that the time-to-peak drug level will be different than with traditional arm freezing procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing brachial plexus anesthesia as part of disease management who have consented to participate in the study

Exclusion Criteria:

* Contraindication to brachial plexus anesthesia
* Informed consent not obtained

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Lidocaine drug level | 40 minutes

SECONDARY OUTCOMES:
brachial plexus block quality | 30 minutes
Physiotherapy quality | within 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric N Sutherland, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Pain Management Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Neal JM, Hebl JR, Gerancher JC, Hogan QH. Brachial plexus anesthesia: essentials of our current understanding. Reg Anesth Pain Med. 2002 Jul-Aug;27(4):402-28. doi: 10.1053/rapm.2002.34377. No abstract available. PMID 12132064
- [Background] Norder H, Hammas B, Larsen J, Skaug K, Magnius LO. Detection of HBV DNA by PCR in serum from an HBsAg negative blood donor implicated in cases of post-transfusion hepatitis B. Arch Virol Suppl. 1992;4:116-8. doi: 10.1007/978-3-7091-5633-9_24. PMID 1450678
- [Background] Soares LG, Brull R, Lai J, Chan VW. Eight ball, corner pocket: the optimal needle position for ultrasound-guided supraclavicular block. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):94-5. doi: 10.1016/j.rapm.2006.10.007. No abstract available. PMID 17196502
- [Background] Beach ML, Sites BD, Gallagher JD. Use of a nerve stimulator does not improve the efficacy of ultrasound-guided supraclavicular nerve blocks. J Clin Anesth. 2006 Dec;18(8):580-4. doi: 10.1016/j.jclinane.2006.03.017. PMID 17175426